CLINICAL TRIAL: NCT06766877
Title: Effect of Core Stability Versus Conventional Exercise for Functional Ambulation of Calf Muscle
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shaikh Nabi Bukhsh Nazir, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMU/Approval?
Record Dates: First submitted 2025-01-02; First posted 2025-01-09 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee; arthritis; tendon
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Core Stability (Experimental): Core Stability exercises:
  Bridging Lateral Step up etc
  Interventions: Other: core stability exercise
- Foot-ankle strengthening exercise (Active Comparator): resistance exercises with proper warm up and cool down
  Interventions: Other: foot-ankle strengthening exercise

INTERVENTIONS:
Other: core stability exercise — 1. Isometric quadriceps exercises involving knee extension
  2. Maximum isometric exercise for the quadriceps
  Arms: Core Stability
Other: foot-ankle strengthening exercise — 1. Isometric quadriceps exercises involving knee extension
  2. Maximum isometric exercise for the quadriceps
  Arms: Foot-ankle strengthening exercise

SUMMARY:
Knee osteoarthritis (KOA) is a degenerative joint disease causing pain, stiffness, and reduced quality of life. While treatments often focus on drugs or surgery, noninvasive exercises like core stabilization and ankle/foot strengthening show potential but lack comparative studies. Understanding anatomical factors like Achilles tendon (AT) thickness is crucial for targeted rehabilitation, though measurement reliability remains an issue. This study aims to compare the effects of these exercises on KOA symptoms and evaluate the use of digital calipers for AT thickness measurement, aiming to enhance clinical management of KOA.

DETAILED DESCRIPTION:
The objective of the study is:

1. To determine the interrater and intrarater reliability of digital calliper to measure the side to side Achilles tendon thickness.
2. To determine the impact of 24 sessions of core stability translated in gait ambulation.
3. determines the relationships between Achilles tendon thickness (ATT), knee symptoms/functions, and foot alignment in knee OA patients, considering their interconnected biomechanical nature.
4. compare the effects of core stability and ankle-foot strengthening exercises on clinical outcomes in KOA patients

ELIGIBILITY:
Inclusion Criteria:

* 40 years old, had been diagnosed with KOA based on ACR, and

  * having Grade II or III osteoarthritis by K/L criteria.

Exclusion Criteria:

* post-traumatic osteoarthritis
* lower limb sensorimotor dysfunction,
* Any history of knee fracture/ tumor/ infection and hip/knee surgery.
* Total Knee Replacement patients.
* Neurological disease.
* Patient received physical therapy treatment from last 6 months.
* Inflammatory Arthritis (Rheumatoid Arthritis)
* Use of any intra-articular injections (steroid/ hyaluronic acid/ PRP.) from last 3-6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-22 (Actual); Primary Completion 2025-02-22 (Estimated); Study Completion 2025-02-23 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) Questionnaire | 8 weeks
  Changes from baseline, KOOS score consist of five patient-relevant dimensions that are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. This scale consist of total 42-items and score of this scale range from 0 (severe knee pathology) to 100 (no knee problem). This tool has been use to assess the pain, symptoms, activities level, function in knee osteoarthritis patients. It is a valid tool for Knee Osteoarthritis patients ; validity ranges up-to (0.80-0.89).
Visual Analogue Scale (VAS) at rest | 8 weeks
  Changes from baseline, Visual Analogue Scale (VAS) is the most commonly used scale in which the pain rate ranges from 0 (no pain) to 10 (worst pain). The level of knee perception of pain is assessed by using the VAS.
Stair climb test | 8 weeks
  change from baseline, time taken to ascend and descend the stairs
Knee flexion range of motion | 8 weeks
  Change from baseline, flexion was assessed with a goniometer
knee extension range of motion | 8 weeks
  change from baseline, extension was assessed with goniometer
Achilles tendon thickness | 8 weeks
  Change from baseline, tendon thickness was measured was assessed with digital calliper
30 second chair test | 8 weeks
  change from baseline, The 30 Second Sit to Stand Test is also known as 30 Second Chair Stand Test (30CST), was initially designed for testing leg strength and endurance in older adults.
Timed up and go test | 8 weeks
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults
40 meter walk test | 8 weeks
  Instruct patient to walk as quickly, but as safely as possible, without running, along 10m walkway, past the taped line, & then turn around cone & return.
Gastrocnemius muscle strength | 8 weeks
  Patient to perform plantar flexion in the form of single-limb heel raise
navicular/foot ratio | 8 weeks
  The midfoot alignment was assessed using the navicular/foot ratio, which is calculated as the ratio of the navicular height to the total foot length.
Ankle range of motion | 8 weeks
  The dorsiflexion range of ankle movement was evaluated using the knee-to-wall lunge technique

CONTACTS AND LOCATIONS:
Overall Officials: SHAIKH NABI BUKHSH NAZIR, PhD Scholar, Principal Investigator — Dow University of Health Sciences/ Baqai Medical University
Locations (1):
- BIPTRM, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No